CLINICAL TRIAL: NCT01726348
Title: A Post-Marketing Surveillance Study on the Safety and Effectiveness of Darunavir on Filipino Patients With Human Immunodeficiency Virus-Type I (HIV-1) Infection
Brief Title: A Study to Assess the Safety and Effectiveness of Darunavir for Treating Human Immunodeficiency Virus-Type I (HIV-1) Infection in Filipino Patients
Status: Withdrawn | Type: Observational
Why Stopped: The company decided to cancel this study in conformity with PH FDA Circular 2013-004
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014686; TMC114HIV4013 (Other: Janssen Pharmaceutica); PRE-PHL-MA1 (Other: Janssen Pharmaceutica); TMC-C-07-PH-007 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Human Immunodeficiency Virus-Type 1
Keywords: Human Immunodeficiency Virus-Type 1; HIV-1; TMC114; Darunavir; Ritonavir; Filipino
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Darunavir: Patients will be taking darunavir as per the dosing regimen given on product insert approved in Philippines.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Darunavir will be administered as per the recommended doses and will be given orally every 4 weeks for a period of 24 weeks. For treatment-naive and treatment-experienced adult patients with no darunavir resistance associated substitutions: Darunavir 800 mg will be administered with ritonavir 100 mg once daily with food. For treatment-experienced adult patients with at least one darunavir resistance associated substitution: Darunavir 600 mg will be administered with ritonavir 200 mg twice daily with food.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of darunavir for the treatment human immunodeficiency virus-type I (HIV-1) infection among Filipino adults.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (study conducted at multiple sites), uncontrolled (all the patients receiving darunavir) clinical and observational study (study in which the investigators/physicians observe the patients and measure their outcomes) to evaluate the safety and effectiveness of darunavir for the treatment human immunodeficiency virus-type 1 (HIV-1) infection among adult Filipino patients. The study will enroll 10 percentage of patient who would use the product, as a requirement of the Philippine Food and Drug Administration (FDA). Patients will be monitored from baseline and every 4 weeks thereafter for a period of 24 weeks. Safety evaluations for adverse events, clinical laboratory tests, physical examination, concomitant medications, and co-morbid conditions will be monitored throughout the study. The duration of treatment will be for 24 weeks and the total study will be conducted for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with human immunodeficiency virus-type 1 (HIV-1), and who are eligible for darunavir (in combination with ritonavir) treatment. These may be either: treatment-naive adult patients and treatment-experienced adult patients with no darunavir resistance associated substitutions; or treatment-experienced adult patients with at least one darunavir resistance associated substitution

Exclusion Criteria:

* Known hypersensitivity to darunavir/ritonavir or to any of the components of the two agent preparations
* Pregnant or breastfeeding females
* Agrees to protocol-defined use of effective contraception
* Patients taking medication that are highly dependent on Cytochrome P450 3A4 for clearance and for which initial concentrations are associated with serious and/or life threatening events
* Patients with severe hepatic impairment
* History of allergy to sulfa containing drugs or molecules
* Patients currently receiving alfuzosin, dihydroergotamine, ergonovine, ergotamine, methylergonavine, cisapride, pimozide, midazolam, triazolam, St. John's Wort (Hypericum perforatum), lovastatin, simvastatin, rifampin and sildenafil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult Filipino patients who are diagnosed with human immunodeficiency virus-type 1 (HIV-1), and who are eligible for darunavir (in combination with ritonavir) treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of adverse events | Up to 24 weeks
Number of patients with incidence of discontinuation of study medication due to adverse events | Up to 24 weeks

SECONDARY OUTCOMES:
Mean decrease of viral load at the end of treatment from baseline | Baseline, Week 12, and Week 24
Number of patients with viral load of 50 copies per ml at the end of treatment | Baseline, Week 12, and Week 24
Number of patients with lack of effect | Up to 24 weeks
  Any failure of expected pharmacologic action of the study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica